CLINICAL TRIAL: NCT04260334
Title: Preoperative Care in Ovarian Cancer: Effects of Relaxation-Focused Nursing Program in Women With Ovarian Cancer
Brief Title: Preoperative Care In Ovarian Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Buse Güler, Research Asisstant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/06-42
Record Dates: First submitted 2019-11-06; First posted 2020-02-07 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Adnexal Mass; Perioperative Complication; Outcome, Fatal
Keywords: Adnexal mass; Preoperative education; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): RFNP was created by researchers. RFNP comprises positive language, a positive environment, relaxation exercise and methods of coping with stress (Mete et al., 2017; Mete et al., 2015; Lazarus, 1984). This programme has a content which reducing women's anxiety and pain. Such programmes are expected to enhanced level of the knowledge about ovarian cancer and its surgery. Women are usually admitted to the clinic two days before surgery. The program duration was for 2 days each day with two sessions, of 6 hr each. There are four relaxation exercises in the program because repetition is recommended for the relaxation exercises to be effective. Deep breathing exercise, progressive muscle relaxation, and guided imagery were used in program. In addition, RFNP is divided into four sections so that the information is not intensely transferred to women.
  Interventions: Other: Preoperative Education
- Control Group (No Intervention): In the control group, women received routine nursing care in the hospital, and data collection tools were applied at the parallel hours as the experimental group. Usual nursing care included information about visitor and meal times, nurse call button, diet, drug administration and not to leave the hospital. Relaxation exercises were not practiced to patients in usual nursing care to reduce stress and anxiety.

INTERVENTIONS:
Other: Preoperative Education — The first two hours after the hospitalization of the patient will be met and the aim of the study will be explained. On the same day, the patient will be given breathing and relaxation exercises and explained why it is important. On the second day after the hospitalization, the patient will be evaluated and the previous day's exercises will be repeated and leg exercises will be performed. The importance of mobilization will then be highlighted. the same day gradual relaxation exercise and surgical relaxation will be administered to the patient three times. The patient will be evaluated on the first postoperative day.
  Arms: Intervention Group

SUMMARY:
A randomised controlled trial study consisting of two-group pretest-post-test.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled trial with pretest and posttest model. The sample of the research consisted of patients who would undergo ovarian cancer surgery at the gynecologic oncology unit of a university hospital in Turkey between June 2019-August 2020.

The women were randomly assigned using "a random number generation program (Research Randomizer (https://www.randomizer.org/)" by an independent researcher who was not included in the study, intervention and control groups were formed. Women were not informed about the group they would be a part of. However, the groups of women were known by the researchers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over
* women who know diagnosis
* women who have not psychiatric illness
* women who have preoperative period
* hospitalization two days before surgery

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Anxiety | 3 days
  It has been measured The State and Trait Anxiety Inventory. Form Y, its most popular version, has 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Scores range from 20 to 80, with higher scores correlating with greater anxiety.
analgesia | 3 days
  It has been measured visual analog scale for pain. Scores range from 0 to 10, with higher scores correlating with greater pain.

CONTACTS AND LOCATIONS:
Overall Officials: Buse Güler, MSc, Principal Investigator — Dokuz Eylul University
Locations (1):
- Health Science University Tepecik Education and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No